CLINICAL TRIAL: NCT05664555
Title: Low Dose Fluorescein Angiography Comparing 1mL and 3mL of 10% Fluorescein: A Randomized Controlled Trial
Brief Title: Dose Optimization for Safe and Efficient Fluorescein Angiography (DOSE Study)
Acronym: DOSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Min Seok Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: B-2211-790-004
Record Dates: First submitted 2022-12-06; First posted 2022-12-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases | interventions — Fluorescein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Na Fluorescein 3mL Arm (Active Comparator): Participants in this arm will receive Na Fluorescein 10% Inj 3mL (300mg) before taking fluorescein angiography.
  Interventions: Drug: Fluorescein Sodium
- Na Fluorescein 1mL Arm (Experimental): Participants in this arm will receive Na Fluorescein 10% Inj 1mL (100mg) before taking fluorescein angiography.
  Interventions: Drug: Fluorescein Sodium

INTERVENTIONS:
Drug: Fluorescein Sodium — Patients will receive Fluorescein Sodium 3mL (300mg) or 1mL (100mg) intravenously prior to fluorescein angiography.

SUMMARY:
This study aims to compare the efficacy and safety of fluorescein angiography using 1mL versus 3mL of 10% fluorescein dye.

DETAILED DESCRIPTION:
The investigators will recruit patients who need fluorescein angiography for their retinal diseases.

The investigators will collect data on image quality and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who required an fluorescein angiography for their retinal diseases (eg. diabetic retinopathy, retinal vein occlusion, etc.)

Exclusion Criteria:

* media opacity (corneal opacity, vitreous hemorrhage grade 2 or more, cataract LOCS III grade 3 or more)
* known history of adverse reactions to fluorescein
* dilated pupil diameter less than 5 mm

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Subjective image quality from 3 experts | One month
  Images from two dose groups will be compared in terms of central and peripheral image quality. Three retinal experts were masked to the fluorescein dose the patients had received. Each expert graded patients' fluorescein angiography images on a scale of 1 to 5 (1:very poor, 2: poor, 3: average, 4: better than average, 5: excellent) with respect to the subjective quality of the image and aid of making a diagnosis. The mean value of the image quality score will be compared between the two dose groups.

SECONDARY OUTCOMES:
Objective vessel intensity | One month
  Mean vascular pixel intensity was quantitatively measured using ImageJ (version 1.54f, National Institutes of Health). The 8-bit grayscale image was imported into imageJ and processed with a top-hat filter to suppress the background noise. This UWFA image was divided via a customized grid, consisting of 2 rings centered on the fovea. The mean vascular pixel intensity in each of these zones was then automatically measured using imageJ software.
Complication | immediately after the test
  frequency of complication of fluorescein angiography will be compared between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Moosbrugger KA, Sheidow TG. Evaluation of the side effects and image quality during fluorescein angiography comparing 2 mL and 5 mL sodium fluorescein. Can J Ophthalmol. 2008 Oct;43(5):571-5. doi: 10.3129/i08-122. PMID 18982034
- [Background] Friberg TR, Gupta A, Yu J, Huang L, Suner I, Puliafito CA, Schwartz SD. Ultrawide angle fluorescein angiographic imaging: a comparison to conventional digital acquisition systems. Ophthalmic Surg Lasers Imaging. 2008 Jul-Aug;39(4):304-11. doi: 10.3928/15428877-20080701-06. PMID 18717436
- [Background] Nasrallah FP, Jalkh AE, Trempe CL, McMeel JW. Low-dose fluorescein angiography. Am J Ophthalmol. 1988 Jun 15;105(6):690. doi: 10.1016/0002-9394(88)90071-2. No abstract available. PMID 3377048
- [Derived] Song SH, Joo K, Woo SJ, Kim MS. IMAGE QUALITY AND SAFETY OF 300 MG VERSUS 100 MG FLUORESCEIN IN ULTRA-WIDEFIELD FLUORESCEIN ANGIOGRAPHY: A Randomized Clinical Trial. Retina. 2025 Jun 1;45(6):1168-1174. doi: 10.1097/IAE.0000000000004420. PMID 39933138